CLINICAL TRIAL: NCT01945138
Title: Efficacy and Feasibility of Fully Automated Closed Loop Insulin Pump Therapy After Islet Auto-Transplantation
Brief Title: Closed Loop Insulin Pump Therapy After Islet Auto-Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLTPIAT2013; 21856 (Other Grant/Funding Number: University of Minnesota - CTSI)
Record Dates: First submitted 2013-08-19; First posted 2013-09-18 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Chronic Pancreatitis; Diabetes Mellitus
Keywords: Total Pancreatectomy; Islet Auto-Transplantation; Closed Loop Insulin Pump
MeSH Terms: conditions — Pancreatitis, Chronic; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control Group: patients receive conventional multiple daily injection insulin therapy with basal and bolus dosing during the 72 hour study period.
- Closed Loop Insulin (Experimental): Closed Loop Insulin Group: patients receive continuous subcutaneous insulin controlled by experimental closed loop system during the 72 hour study period.
  Interventions: Device: Closed Loop Insulin

INTERVENTIONS:
Device: Closed Loop Insulin — The Closed Loop Insulin system is an automated insulin delivery system based on body blood glucose. It consists of an Insulin pump, continuous glucose monitor, and a control device (laptop with algorithms).
  Other Names: Medtronic ePID 2.0 system; Medtronic Paradigm REAL-Time Insulin Pump (MMT-722); Enlite Glucose Sensor (MMT-7008X); MiniLink REAL-Time Transmitter (MMT-7703XNA); ComLink Device (MMT-7304)
  Arms: Closed Loop Insulin

SUMMARY:
The purpose of this study is to determine the effectiveness of closed loop insulin pump therapy to control blood sugar following total pancreatectomy and islet auto-transplantation (TPIAT).

DETAILED DESCRIPTION:
OBJECTIVES AND HYPOTHESES The main objective of this study is to determine if a closed loop insulin system can successfully achieve tighter blood sugar control than the current multiple daily injection regimen. The investigators hypothesize that the average blood glucose will be lower in the closed loop group than the control group, there will be less glucose variability in the closed loop group than the control group, and there will be less total time spent in hyperglycemia and hypoglycemia in the closed loop group than in the control group. The investigators also will investigate insulin requirements and islet function in the first 6 months post-transplant in the closed loop group The investigators hypothesize that the insulin requirements will be lower and the C-peptide levels higher in the closed loop group than in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total pancreatectomy and islet auto-transplantation.
* Patients ages 21 to 64 years old

Exclusion Criteria:

* Preexisting diabetes
* Use of acetaminophen during study period, which interferes with CGM sensor function
* Any medical condition requiring corticosteroids
* Severe Psychiatric disease or developmental delays, that might interfere with the ability to provide informed consent
* Any other medical condition which in the opinion of the investigators impairs the person's ability to safely participate in the trial

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melena Bellin, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Forlenza GP, Nathan BM, Moran AM, Dunn TB, Beilman GJ, Pruett TL, Bellin MD. Successful Application of Closed-Loop Artificial Pancreas Therapy After Islet Autotransplantation. Am J Transplant. 2016 Feb;16(2):527-34. doi: 10.1111/ajt.13539. Epub 2015 Nov 20. PMID 26588810

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Closed Loop Insulin
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Closed Loop Insulin | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (13.3) | 38.6 (9.4) | 35.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 4 | 1 | 5
Weight at Transplant [Mean (Standard Deviation); unit: kg] | 76.7 (23.7) | 66.1 (10.3) | 71.4 (18.4)
Body Mass Index (BMI) at Transplant [Mean (Standard Deviation); unit: kg/m2] | 24.9 (5.7) | 25.3 (4.5) | 25.1 (4.9)
hemoglobin A1c (A1c) [Mean (Standard Deviation); unit: %] | 5.4 (0.5) | 5.1 (0.2) | 5.3 (0.4)
Fasting Blood Glucose (BG) [Mean (Standard Deviation); unit: mg/dL] | 95 (13) | 89 (6) | 92 (10.3)
Fasting C-Peptide [Mean (Standard Deviation); unit: ng/mL] | 95 (13) | 89 (6) | 92 (10.3)
Peak Mixed Meal Tolerance Test (MMTT) C-peptide [Mean (Standard Deviation); unit: ng/mL] | 5.8 (4.4) | 6.4 (2.2) | 6.1 (3.4)
Islet Yield [Mean (Standard Deviation); unit: IEq/kg] | 4245 (2174) | 6619 (3357) | 5432 (2983)
Days on drip [Mean (Standard Deviation); unit: days] | 6.9 (1.1) | 5.1 (1.1) | 6.0 (1.4)
Etiology of Chronic Pancreatitis (CP) [Number; unit: participants]
  Identified Genetic Mutation (PRSS1, SPINK1, CFTR) | 1 | 3 | 4
  Mechanical Dysfunction | 4 | 3 | 7
  Idiopathic Pancreatitis | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Study Period: Average Serum BG
Description: Mean blood glucose value: a single report of the average of the analytical blood glucose values will be computed and compared between the pump and control groups.
Time Frame: 3 days of investigation period
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
mg/dL | 130 (13) | 111 (4)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

2. Primary Outcome: Study Period: Serum BG Standard Deviation
Description: Measure of glycemic variability. This is the standard deviation in all serum BG values for each individual patient.
Time Frame: 3 days of investigation period
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
mg/dL | 21.0 (10.2) | 14.1 (3.3)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.115, t-test, 2 sided

3. Secondary Outcome: Study Period: Continuous Glucose Monitor (CGM) BG Average
Description: Continuous glucose monitoring sensor data: The CGM's in the pump and control groups will collect glucose readings continuously over a 72 hour period
Time Frame: continuously over the 72 hour investigational period
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
mg/dL | 125 (20) | 114 (4)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.193, t-test, 2 sided

4. Secondary Outcome: Study Period: Continuous Glucose Monitor Standard Deviation of BG
Description: measure of glycemic variability by CGM. This is the standard deviation within each patient for all CGM glucose readings.
Time Frame: continuous over the 72 hour investigation period
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
mg/dL | 21.0 (10.3) | 20.1 (5.1)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.848, t-test, 2 sided

5. Secondary Outcome: Study Period: Percent Time BG in Range 70-140 mg/dL
Description: Additional measure of glycemic variability, as reflected by CGM measures, % time in the range of 70-140 on CGM
Time Frame: continuous over the 72 hour investigation period
Measure: Mean (95% Confidence Interval); unit: % of time
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
% of time | 70.6 [48.0 to 93.1] | 89.2 [83.5 to 94.8]
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.074, t-test, 2 sided

6. Secondary Outcome: Study Period: CGM Area Under the Curve (AUC) With Glucose < 70 mg/dL
Description: Calculated as the area under the curve on the CGM tracing that the glucose is under 70 mg/dL.
Time Frame: continuous over the 72 hour investigation period
Measure: Mean (Standard Deviation); unit: min*mg/dL/day
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
min*mg/dL/day | 1615 (4267) | 146 (270)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.38, t-test, 2 sided

7. Secondary Outcome: Study Period: % of Time CGM BG <70 mg/dL
Time Frame: continuous over the 72 hour investigation period
Measure: Mean (95% Confidence Interval); unit: % of time
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
% of time | 4.8 [-6.9 to 16.6] | 1.1 [-0.3 to 2.6]
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.461, t-test, 2 sided

8. Secondary Outcome: Study Period: CGM AUC With Glucose> 140 mg/dL
Time Frame: continuous over the 72 hour investigation period
Measure: Mean (Standard Deviation); unit: min*mg/dL/day
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
min*mg/dL/day | 7860 (11444) | 2025 (1177)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.205, t-test, 2 sided

9. Secondary Outcome: Study Period: % of Time CGM BG > 140 mg/dL
Time Frame: continuous over the 72 hour investigation period
Measure: Mean (95% Confidence Interval); unit: % of time
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
% of time | 23.7 [1.5 to 46.0] | 9.7 [4.9 to 14.5]
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.157, t-test, 2 sided

10. Secondary Outcome: Study Period: Morning C-peptide
Description: A single C-peptide measurement collected daily x 3 days, collected at random (meaning not in a fasting state) each morning. Expressed as average for each patient.
Time Frame: Average of 3 day study period
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
ng/mL | 1.6 (1.0) | 1.3 (0.6)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.443, t-test, 2 sided

11. Secondary Outcome: Study Period: Daily Insulin Needs
Description: Calculated as total daily dose of insulin.
Time Frame: Average of 3 day study period
Measure: Mean (Standard Deviation); unit: U/kg/day
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
U/kg/day | 0.56 (0.31) | 0.26 (0.17)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

12. Secondary Outcome: Day 14 Follow-Up: Average Serum BG
Time Frame: Day 14 Follow-Up
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
mg/dL | 135 (81) | 106 (16)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.401, t-test, 2 sided

13. Secondary Outcome: Day 14 Follow-Up: C-Peptide
Time Frame: Day 14 Follow-Up:
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
ng/mL | 1.0 (0.9) | 1.6 (0.9)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.22, t-test, 2 sided

14. Secondary Outcome: Day 28 Follow-Up: Average Serum BG
Time Frame: Day 28 Follow-Up
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
mg/dL | 113 (29) | 100 (21)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.325, t-test, 2 sided

15. Secondary Outcome: Day 28 Follow-Up: C-Peptide
Time Frame: Day 28 Follow-Up
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Control | Closed Loop Insulin
Number analyzed (Participants) | 7 | 7
ng/mL | 1.0 (1.2) | 1.7 (1.2)
Statistical Analysis 1: Comparison: Control vs Closed Loop Insulin; Test type: Superiority or Other; p = 0.311, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Control | Closed Loop Insulin
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 2/7 | 3/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=7) | Closed Loop Insulin (N=7)
Mild Hypoglycemia (Endocrine disorders) | 1 (2) | 3 (3)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes